CLINICAL TRIAL: NCT04218214
Title: LIFE-DM Implementation Study: A Mixed Methods Implementation Evaluation of an Integrated Depression and Microfinance Program for Women in Vietnam
Brief Title: Mixed Methods Implementation Evaluation of an Integrated Depression and Microfinance Program for Women in Vietnam
Acronym: LIFE-DM
Status: Completed | Type: Observational
Sponsor: RAND (Other)
Collaborators: Grand Challenges Canada (Other); Basic Needs Vietnam (Unknown); Danang Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Victoria K. Ngo, PhD, Principal Investigator, RAND
Other Study IDs: 2017-0716
Record Dates: First submitted 2018-05-11; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: depression; poverty
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LIFE-DM Group: The LIFE-DM group is a 12-session based on Behavior Activation and Problem Solving therapy for depression applied to both mood problems and livelihood stressors. Livelihood supports includes training on personal finance, referrals to vocational training, and microfinance loans of 2 million VND. The group is provided at the local commune health stations, and facilitated by primary care health provider and a lay community provider from the Women's Union.
  Interventions: Other: LIFE-DM Group (Integrated Depression and Livelihood Group Intervention)

INTERVENTIONS:
Other: LIFE-DM Group (Integrated Depression and Livelihood Group Intervention) — Livelihood Integration for Effective Depression Management (LIFE-DM) program aims to address the dual challenges of poverty and depression by integrating evidence-based treatment for depression management and microfinance services. The LIFE-DM group is a 12-session based on Behavior Activation and Problem Solving therapy for depression applied to both mood problems and livelihood stressors. Livelihood supports includes training on personal finance, referrals to vocational training, and access to microfinance loans. The group is provided at the local commune health stations, and facilitated by primary care health provider and a lay community provider from the Women's Union. The intervention generally lasts about 3-4 months.
  Other Names: Livelihood Integration for Effective Depression Management; behavior activation; problem solving; microfinance

SUMMARY:
This is an implementation project to develop a model to support implementation of LIFE-DM, an evidence-based practice (EBP) program that integrates depression management with microfinance services to address both poverty and depression among low-income women in Vietnam. This evaluation is a mixed methods study that will 1) describe the development of community-partnered implementation process, 2) study the effectiveness of the training and implementation support plan on provider and patient outcomes, and 3) identify factors that impact implementation success.

DETAILED DESCRIPTION:
Livelihood Integration for Effective Depression Management (LIFE-DM) aims to address the dual challenges of poverty and depression faced by women in Vietnam by integrating evidence-based treatment for depression management and microfinance services. With funding from NIMH, the investigators established initial evidence for the effectiveness of LIFE-DM in reducing depression and improving functioning, social support, self-efficacy, and income at six months. These treatment effects were maintained at twelve months, suggesting that the LIFE-DM program may be an effective strategy to break the cycle of depression and poverty in low-income women.

For the Grand Challenges of Canada (GCC) Transition to Scale Grant, the investigators developed a model to scale up the program in the public health and social system across two provinces, Danang and Thua Thien Hue through 1) the training of local trainers from the psychiatric hospital to support local implementation, 2) development of a supervision model, and 3) use of a learning collaborative.

To evaluate the success of the model, the investigators will conduct a mixed methods implementation study that will assess implementation and patient outcomes according to the RE-AIM framework, as well as identify barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* depression - based on Patient Health Questionnaire Total Score = > 9
* low-income
* female
* ages 18 - 60

Exclusion Criteria:

* psychosis risk
* mania risk
* substance abuse risk
* high suicide risk
* physical disabilities
* significant cognitive impairments

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Study participants are recruited from community health clinics that are implementing LIFE-DM and depression care services in the GCC funded transition to scale grant. These participants are 18-60 years old, have elevated depressive symptoms (PHQ 9 > 9), have economic disadvantage, and are interested in participating in an integrated depression and livelihood program. Patients with severe mental illness, such as psychosis, mania, substance abuse, or high risk of suicide are also excluded and referred to psychiatric hospital for higher level of care. Those who have disabilities, significant cognitive impairments, and chronic illness that may interfere with their ability to participate in group therapy are also excluded and referred to other more individualized support.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Provider Adoption of LIFE-DM and Depression Care - Count | one year
  Delivery of LIFE-DM and depression care components (Counts of depression care components delivered - # of screening, assessment, LIFEDM, individual therapy, medication, loans)
Provider Adoption of LIFE-DM and Depression Care - Percentage | one year
  Delivery of LIFE-DM and depression care components (% of depression care components delivered - screening, assessment, LIFEDM, individual therapy, medication, loans based on eligible cases)
Patient Depression Scores (PHQ) Change from Baseline to 6 month | 0, 6 months
  Patients will be assessed for depression using self-reported depression measure (PHQ). The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total scores are used and they range from 0 to 27, with PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Provider Participation | 0-12 months
  Provider Participation in Training Activities (Count / % of workshop attendance, supervision meetings, and learning collaborative meetings)
Provider Implementation Quality | throughout the study implementation period, about 1 year
  Supervisor Rated LIFE-DM session adherence and quality. Supervision of groups involve observation of group facilitation by supervisors, who provide adherence and quality ratings of sessions. Each item is assessed on a 4 point scale - 0 (did not do), 1 (delivered but poor), 2 (average), and 3 (excellent). The items are averaged to provide a session specific score of adherence and quality. Session adherence / quality scores are used to compute provider level adherence and quality averages. Each supervisor was expected to provide ratings for a minimum of 3 assessments out of the 12 group sessions. These session ratings are used to compute the average adherence and quality score for each provider.
Implementation Barriers and Facilitators | one year
  Qualitative Interviews of Providers and Program Staff to Assess Barriers and Facilitators of Implementation
Change in Patient Functioning | 0 and 6 months
  Patient - SF-12 - Change in functioning from baseline to 6 months. The SF-12 Health Survey is a 12-item subset of the SF-36v2™ that measures the same eight domains of health (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health). It is a brief, reliable measure of overall health status. Scores are calibrated so that 50 is the average score or norm. This norm-based score allows comparison among the three surveys and across the more than 19,000 studies published in the past 20 years
Change in Patient Family Functioning | 0 and 6 months
  Patient - McMaster Family Functioning Scale - Change from baseline to 6 months. This is a 12 item scale (on a 4 point scale). the average score across items is used to determine the degree of problematic family functioning. A score of 2.00 or above indicates problematic family functioning. The higher the score, the more problematic the family member perceives the family's overall functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ngo, PhD, Principal Investigator — RAND
Locations (2):
- Vietnam (2):
  - Commune Health Stations, Huế, Thừa Thiên Huế Province
  - Commune Health Stations, Da Nang

IPD SHARING:
Plan to Share IPD: No